CLINICAL TRIAL: NCT00366665
Title: Comparison of the Infiniti Vision and the Series 20000 Legacy Systems
Brief Title: Comparison of the Performance of the Infiniti Vision and the Series 20000 Legacy Phacoemulsification Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MRC-05-002
Record Dates: First submitted 2006-08-17; First posted 2006-08-21 (Estimated); Last update posted 2006-08-21 (Estimated); Status verified 2005-05

CONDITIONS: Cataract Extraction

INTERVENTIONS:
Device: Legacy 20000
Device: Infinit system

SUMMARY:
To compare the efficiency of the Infiniti vision system and the Series 20000 Legacy System phacoemulsification units during routine cataract extraction.

ELIGIBILITY:
Inclusion Criteria:

* Cataract
* Eligible for cataract extraction with primary implantation of a posterior chamber IOL
* 2 to 3+ cataract density

Exclusion Criteria:

* Preoperative ocular pathology that can affect visual acuity
* Corneal irregularities such as keratoconus, corneal dystrophy, corneal opacities.
* Previous intraocular or corneal surgery.
* Other ocular surgery at the time of the cataract extraction.
* Surgical Exclusion Criteria:
* Significant intraoperative intraocular bleeding
* Detached Descemet's membrane
* Implantation of the intraocular lens in the anterior chamber or sulcus

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-03; Study Completion 2005-05

PRIMARY OUTCOMES:
Ultrasound time
Amount of fluid used
Post operative visual acuity.

CONTACTS AND LOCATIONS:
Overall Officials: Kerry D. Solomon, MD, Principal Investigator — Medical University of South Carolina